CLINICAL TRIAL: NCT04412889
Title: A Study of B-Cell Maturation Antigen/Cluster of Differentiation 19 Dual-Target Chimeric Antigen Receptor T Cell Immunotherapy for Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of BCMA/CD19 Dual-Target CAR-T Cell Immunotherapy for Relapsed or Refractory MM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: Gracell Biotechnology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGC010
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): The patients will receive BCMA/CD19 dual-target CAR-T cell treatment. BCMA/CD19 dual-target CAR-T cell dosage ranges from 2×10^5 to 1×10^6 CAR+T/Kg.
  Interventions: Biological: BCMA/CD19 dual-target CAR-T cell immunotherapy

INTERVENTIONS:
Biological: BCMA/CD19 dual-target CAR-T cell immunotherapy — The intervention is a CAR-T cell immunotherapy targeted CD19 and BCMA. The dosage ranges from 2×10^5 to 1×10^6 CAR+T/Kg.

SUMMARY:
The study is an early, open, single-centered trial. The aim of this study is to evaluate the safety and tolerance of BCMA/CD19 dual-target CAR-T cell immunotherapy in relapsed or refractory MM. The study will include 18 subjects to receive BCMA/CD19 dual-target CAR-T cell immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Diagnosis of relapsed or refractory multiple myeloma (MM): 1) Received at least 3 prior lines of treatment, including proteasome inhibitor (such as bortezomib and carfilzomib) and immunomodulator (such as lenalidomide and pomalidomide), and undergone at least 1 complete cycle of treatment for each line, unless PD was documented as the best response to the regimen; 2) Resistant to proteasome inhibitor and immunomodulator, PD in 60 days after treatment;
3. Measurable disease at screening as defined by any of the following: 1) Serum monoclonal paraprotein (M-protein) level ≥10 g/L or urine M-protein level ≥200 mg/24 hours or; 2) Light chain MM without measurable disease in the serum or the urine: serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa/lambda free light chain ratio or; 3) Plasma cell percentage in bone marrow ≥30%;
4. Histologically confirmed positive expression of CD19 and/or BCMA ≤3 months prior to enrollment;
5. Eastern cooperative oncology group (ECOG) performance status of 0 to 1;
6. Life expectancy≥12 weeks;
7. Adequate organ function is defined as: 1) Hemoglobin≥6.0g/dL (did not receive red blood cell transfusion ≤7 days prior to laboratory tests); 2) Platelet count >50×10^9/L (did not receive blood transfusion ≤7 days prior to laboratory tests); 3) Absolute neutrophil count (ANC) ≥0.75×10^9/L (did not receive supportive treatment ≤7 days prior to laboratory tests); 4) Bilirubin <2×ULN, expect for subjects with congenital hyperbilirubinemia (for subjects with Gilbert's syndrome, direct bilirubin≤2×ULN); 5) Creatinine clearance (according to modification of diet in renal disease formulas or 24h urine collection result) ≥40 mL/min/1.73m^2; 6) Alanine aminotransferase/aspartate aminotransferase (ALT/AST) <2.5×ULN; 7) Corrected serum calcium ≤14 mg/dL (≤3.5 mmol/L), or free calcium ion ≤6.5 mg/dL (≤1.6 mmol/L); 8) Oxygen saturation >92% on non-oxygen-therapy state; 9) Left ventricular ejection fraction (LVEF)>50%, no evidence of clinically significant pericardial effusion as determined by an echocardiography;
8. Meet the requirements of peripheral blood mononuclear cells (PBMC) collection of the site;
9. Females must not be in pregnancy nor in lactation. Form signing the ICF to the end of the trial, females of childbearing potential and males must use efficient contraception;
10. Sign the informed consent form (ICF), can understand and adhere to the procedures and requirements in this study.

Exclusion Criteria:

1. Solitary plasmacytoma;
2. Central nervous system (CNS) involvement;
3. Previous other CAR-T or other gene-editing T cell therapy ≤8 weeks prior to enrollment (not applicable to subject received CAR-T second infusion);
4. Previous allogeneic stem cell transplant; previous autologous stem cell transplant ≤12 weeks prior to enrollment;
5. Any result of the following virology tests is positive: HIV；HCV；HBsAg；HBcAg；TPPA;
6. Concomitant malignancy that require treatment or do not achieve complete remission in 3 years prior to enrollment other than: cured non-melanoma skin cancer, cervical carcinoma in situ, prostate cancer that do not require treatment, other malignancy whose disease-free survival exceeds 5 years;
7. Toxicities related to previous therapy did not relieved to ≤1 grade, except hematological toxicity and alopecia;
8. Live vaccine ≤4 weeks prior to enrollment;
9. Other investigational drug ≤4 weeks prior to enrollment;
10. Surgical operation that require general anesthesia happened ≤4 weeks prior to enrollment, or did not be fully recovered and clinically stable prior to enrollment, or be anticipated to undergo major surgical operation that require general anesthesia during the study;
11. Any unstable cardiovascular disease happened ≤6 months prior to enrollment, including but not limited to, unstable angina, myocardial infarction, heart failure (NYHA grade ≥ III grade), severe arrhythmia that require drug interference, cardiac angioplasty/coronary stent implantation/cardiac bypass surgery ≤6 months prior to enrollment;
12. Presence of active autoimmune disease (including but not limited to, systemic lupus erythematosus, sjogren syndrome, rheumatoid arthritis, inflammatory bowel disease, hypothyroidism which can be controlled by thyroid hormone replacement therapy is an exception);
13. Presence of CNS disease or disease history, including epilepsy, cerebral ischemia/bleeding, dementia, cerebellar disease (not applicable to subject received CAR-T second infusion, unless 4 grade ICANS happened after CAR-T first infusion);
14. Presence of complication that require systemic corticosteroids or other immunosuppressive drugs therapy during the trial in researcher's judgement;
15. Known life-threatening hypersensitivity to cyclophosphamide or fludarabine, or presence of other intolerant conditions, or severe allergic constitution;
16. Presence of plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome or primary amyloidosis;
17. Any other condition that researcher think it is inappropriate for the subject to anticipate the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Type and incidence of dose-limiting toxicity (DLT), incidence and severity of treatment related adverse event (AE), cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome, ICANS) (safety and tolerability) | 2 years
  AE will be collected and graded according to American Society for Transplantation and Cellular Therapy (ASTCT) consensus (for CRS/ICANS) and CTCAE v5.0(for AE except CRS/ICANS)

SECONDARY OUTCOMES:
CAR copies in peripheral blood, bone marrow, extramedullary plasmacytoma, and cerebrospinal fluid (CSF) (amplification and persistence) | 2 years
  CAR copies in peripheral blood, bone marrow, extramedullary plasmacytoma and CSF will be measured by quantitative polymerase chain reaction (qPCR) in 2 years.
CAR cells in peripheral blood, bone marrow and CSF (amplification and persistence) | 2 years
  CAR cells in peripheral blood, bone marrow and CSF will be measured by flow cytometry (FCM) in 2 years.
Objective response rate (ORR) (efficacy) | 6 months
  ORR will be calculated as the percentage of patients who achieved partial response (PR) or better.
Duration of response (DOR) (efficacy) | 2 years
  DOR will be calculated as the time from the first assessment of PR or better to the first assessment of progressive disease (PD) or death from any cause.
Progression-free survival (PFS)(efficacy) | 2 years
  PFS will be calculated as the time from CAR-T infusion to disease progression or death from any cause (whichever occurs first).
Overall survival (OS)(efficacy) | 2 years
  OS will be calculated as the time from CAR-T infusion to death from any cause.
Concentration of anti-CAR antibody after infusion (humoral immune response) | 2 years
  After CAR-T infusion, anti-CAR antibody in peripheral blood will be measured in 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China